CLINICAL TRIAL: NCT02962011
Title: Randomized Trial Comparing Barbed and Non-barbed Suture for Uterine Incision Closure at Cesarean Section
Brief Title: Trial Comparing Barbed and Non-barbed Suture for Uterine Incision Closure at Cesarean Section
Acronym: barbed
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, David Peleg, MD, Ziv Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZIVH
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Cesarean Section
Keywords: Cesarean, incision, suture,
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Intervention Model Description: Knotless barbed suture vs conventional suture of uterine incision
Who Masked: Participant
Masking Description: unblinded
Oversight: Data Monitoring Committee: No

ARMS (2):
- Knotless barbed suture (Experimental)
  Interventions: Device: Knotless barbed suture
- polyglactin 910 (Active Comparator): Vicryl
  Interventions: Device: polyglactin 910

INTERVENTIONS:
Device: Knotless barbed suture — uterine incision closure
  Other Names: Stratafix
  Arms: Knotless barbed suture
Device: polyglactin 910 — uterine incision closure
  Other Names: Vicryl
  Arms: polyglactin 910

SUMMARY:
This was an unblinded randomized controlled trial. Women were randomized to uterine closure with the knotless barbed suture (Stratafix PDS, Ethicon) or Vicryl (Ethicon) at the time of elective cesarean. The primary outcome was closure time of the uterine incision. Also measured were blood loss during incision closure and the use of additional hemostatic sutures. Informed consent was obtained

ELIGIBILITY:
Inclusion Criteria:

* elective cesarean
* elective repeat cesarean

Exclusion Criteria:

* emergent or urgent cesarean
* PROM
* chorioamninitis
* placental abruption
* placenta previa or accreta
* known uterine fibroids
* women with known medical problems such as coagulopathy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Uterine incision closure time | 5 months
  uterine incision closure time

SECONDARY OUTCOMES:
uterine incision blood loss | 5 months
  uterine incision blood loss
hemostatic suture use | 5 months
  hemostatic suture use

CONTACTS AND LOCATIONS:
Overall Officials: David Peleg, Principal Investigator — Ziv Medical Center
Locations (1):
- Ziv Medical Center, Safed, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peleg D, Ahmad RS, Warsof SL, Marcus-Braun N, Sciaky-Tamir Y, Ben Shachar I. A randomized clinical trial of knotless barbed suture vs conventional suture for closure of the uterine incision at cesarean delivery. Am J Obstet Gynecol. 2018 Mar;218(3):343.e1-343.e7. doi: 10.1016/j.ajog.2018.01.043. Epub 2018 Feb 5. PMID 29496259